CLINICAL TRIAL: NCT03217253
Title: A Phase I Study of Single Agent Tazemetostat in Subjects With Advanced Solid Tumors and B-Cell Lymphomas With Hepatic Dysfunction
Brief Title: Tazemetostat in Treating Patients With Metastatic or Unresectable Solid Tumors or B-Cell Lymphomas With Liver Dysfunction
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Other - Drug Manufacturer decision to close study
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2017-01231; NCI-2017-01231 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PJC-025; 10130 (Other: University Health Network Princess Margaret Cancer Center LAO); 10130 (Other: CTEP); UM1CA186644 (NIH)
Record Dates: First submitted 2017-07-12; First posted 2017-07-14 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-01

CONDITIONS: Ann Arbor Stage III B-Cell Non-Hodgkin Lymphoma; Ann Arbor Stage IV B-Cell Non-Hodgkin Lymphoma; Metastatic Malignant Solid Neoplasm; Stage III Hepatocellular Carcinoma AJCC v7; Stage IIIA Hepatocellular Carcinoma AJCC v7; Stage IIIB Hepatocellular Carcinoma AJCC v7; Stage IIIC Hepatocellular Carcinoma AJCC v7; Stage IV Hepatocellular Carcinoma AJCC v7; Stage IVA Hepatocellular Carcinoma AJCC v7; Stage IVB Hepatocellular Carcinoma AJCC v7; Unresectable Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis; Carcinoma, Hepatocellular | interventions — tazemetostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (tazemetostat) (Experimental): Patients receive tazemetostat PO BID on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Tazemetostat

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Tazemetostat — Given PO
  Other Names: E7438; EPZ-6438; EPZ6438

SUMMARY:
This phase I trial studies the best dose and side effects of tazemetostat in treating patients with solid tumors or B-cell lymphomas with liver dysfunction that have spread to other places in the body or cannot be removed by surgery. Tazemetostat may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine safety, tolerability and recommended phase 2 dose (RP2D) of tazemetostat in patients with varying degrees of hepatic dysfunction.

SECONDARY OBJECTIVES:

I. To assess the pharmacokinetics (PK) profiles of tazemetostat in patients with varying degrees of hepatic dysfunction.

II. To observe preliminary antitumor activity of tazemetostat in this population, especially in tumors with aberrations in EZH2 or SWI/SNF complex pathways.

OUTLINE: This is a dose escalation study.

Patients receive tazemetostat orally (PO) twice daily (BID) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically and/or cytologically confirmed solid tumors or B cell lymphoma that are metastatic or unresectable and for which standard treatment options do not exist; patients with hepatocellular carcinoma are eligible without pathological diagnosis if diagnosed on the basis of blood work and imaging
* Patients with evaluable disease will be eligible
* All patients must have completed any prior chemotherapy, targeted therapy and major surgery, >= 28 days before study entry; for daily or weekly chemotherapy without the potential for delayed toxicity, a washout period of 14 days may be acceptable, and questions related to this can be discussed with study principal investigator
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy of greater than 3 months
* Able to swallow and retain orally-administered medication and does not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels
* All prior treatment-related toxicities must be Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 grade =< 1 (except alopecia) at the time of enrollment
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 90 g/L (9.0 g/dL)
* Creatinine within normal institutional limits OR calculated creatinine clearance >= 60 mL/min/1.73 m^2 (Cockcroft-Gault formula) for patients with creatinine levels above institutional normal
* Patients with abnormal hepatic function will be eligible and will be grouped according to criteria; patients with active hemolysis should be excluded; no distinction should be made between liver dysfunction due to metastases and liver dysfunction due to other causes; this data will be captured in the case report form (CRF); registration laboratory investigations will be used to assign a patient to a hepatic function group; hepatic function tests should be repeated within 24 hours prior to starting initial therapy and may result in patients' group assignment being altered if different to registration test results
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of < 1% per year during the treatment period and for 30 days after tazemetostat discontinuation

  * A woman is considered to be of childbearing potential if she is postmenarchal, has not reached a postmenopausal state (>= 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus)
  * Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, established, proper use of hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices
  * Female subjects who use hormonal contraceptives should use an additional barrier method of birth control while on study treatment and for 30 days after discontinuation of study treatment
  * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical study and the preferred and usual lifestyle of the patient; periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures and agreement to refrain from donating sperm, as defined below:

  * With female partners of childbearing potential or pregnant female partners, men must remain abstinent or use a condom during the treatment period and for at least 4 months after the last dose of study drug; men must refrain from donating sperm during this same period; in addition, female partners of male subjects should adhere to the following:

    * Intrauterine device (IUD)(must provide medical documentation of IUD)
    * Hormonal contraceptive (partner must be on a stable dose of the same hormonal contraceptive product for at least 4 weeks before receiving study drug) AND a condom (hormonal contraceptives must be supplemented with condoms)
  * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical study and the preferred and usual lifestyle of the patient; periodic abstinence and withdrawal are not acceptable methods of contraception
* Females of childbearing potential must have a negative serum pregnancy test at screening
* Ability to understand and the willingness to sign a written informed consent document
* Has a QT interval corrected by Fridericia's formula (QTcF) =< 450 msec
* Whenever available, archival tissue (block or minimum 10 slides) is requested for molecular characterization, e.g. detection of somatic mutations and/or candidate biomarkers of response; this is not mandatory and lack of available tissue would not be an exclusion criteria

Exclusion Criteria:

* Symptomatic or untreated leptomeningeal or brain metastases or spinal cord compression as documented by computed tomography (CT) or magnetic resonance imaging (MRI) scan, analysis of cerebrospinal fluid or neurological exam; patients with primary glioblastoma multiforme are excluded
* Radiation therapy in the last 14 days; palliative radiation to a localized area without residual toxicity requires a washout of greater than 7 days
* Clinically significant bleeding diathesis or coagulopathy, including known platelet function disorders; patients on anticoagulation with low molecular weight heparin are allowed
* Known hypersensitivity to any of the components of tazemetostat
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to tazemetostat
* Concurrent investigational agent or anticancer therapy

  * Note: megestrol [Megace] if used as an appetite stimulant is allowed
  * Concurrent treatment with bisphosphonates is permitted; however, treatment must be initiated prior to the first dose of study therapy; prophylactic use of bisphosphonates in patients without bone disease is not permitted, except for the treatment of osteoporosis
  * The concurrent use of all herbal supplements is prohibited during the study (including, but not limited to, St. John's wort, kava, ephedra [ma huang], ginkgo biloba, dehydroepiandrosterone [DHEA], yohimbe, saw palmetto, or ginseng)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, clinically significant bleeding diathesis or coagulopathy, including known platelet function disorders, symptomatic congestive heart failure, unstable angina pectoris, clinically significant cardiac arrhythmias, or psychiatric illness/social situations that would limit compliance with study requirements
* Active hepatitis B virus (HBV; hepatitis B surface antigen [HepBsAG] positive [+ve] and IgM anti-hepatitis B virus core antibody [HBc]), or hepatitis C virus (HCV; detectable HCV ribonucleic acid [RNA]) infection; patients with chronic or cleared HBV and HCV infection are eligible
* Patients with known human immunodeficiency virus (HIV) infection are eligible if being treated with non-interacting antiretroviral (ARV) agents or be willing to stop ARV for the protocol
* Treatment with strong inhibitors or inducers of CYP3A are prohibited from 14 days prior to the first dose of tazemetostat to the end of the study
* Active gastrointestinal tract disease with malabsorption syndrome or unable to swallow oral medications
* Any condition or medical problem in addition to the underlying malignancy and organ dysfunction that the investigator feels would pose unacceptable risk
* Has thrombocytopenia, neutropenia, or anemia of grade >= 3 (per CTCAE 5.0 criteria) or any prior history of myeloid malignancies, including myelodysplastic syndrome (MDS)
* Has abnormalities known to be associated with MDS (e.g. del 5q, chr 7 abn) and multiple primary neoplasms (MPN) (e.g. JAK2 V617F) observed in cytogenetic testing and DNA sequencing
* Has a prior history of T-acute lymphoblastic lymphoma (T-LBL)/T-acute lymphoblastic leukemia (ALL)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2019-09-19 (Actual); Study Completion 2019-09-19 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events of tazemetostat in patients with varying degrees of hepatic dysfunction assessed using Common Terminology Criteria for Adverse Events version 5.0 | Up to 2 years
  Frequency and severity of adverse events will be tabulated using counts and proportions detailing frequently occurring, serious and severe events of interest. Adverse events will be summarized using all adverse events experienced, although a sub-analysis may be conducted including only those adverse events in which the treating physician deems possibly, probably or definitely attributable to study treatment.
Recommended phase 2 dose (RP2D) of tazemetostat in patients with varying degrees of hepatic dysfunction | Up to 2 years
  RP2D will be determined.

SECONDARY OUTCOMES:
Pharmacokinetic (PK) profiles of tazemetostat in patients with varying degrees of hepatic dysfunction | Up to course 4 day 1 (day 85)
  Plasma concentrations will be measured by Q2 Solutions using a validated Liquid chromatography (LC)/mass spectrometry (MS)/MS assay. Molecular and clinical predictors of clinical outcomes will be investigated using logistic regression and Cox proportional hazards models. Potential predictors include clinical predictors and molecular correlates. Descriptive statistics and plotting of data will also be used to better understand potential relationships. Given the small sample size, and exploratory nature of these endpoints, all pharmacodynamic analyses conducted will be considered exploratory. All analyses will be considered exploratory and inference will be performed with appropriate caution.
Antitumor activity of tazemetostat | Up to 2 years
  Molecular and clinical predictors of clinical outcomes will be investigated using logistic regression and Cox proportional hazards models. Potential predictors include clinical predictors and molecular correlates. Descriptive statistics and plotting of data will also be used to better understand potential relationships. All analyses will be considered exploratory and inference will be performed with appropriate caution.
Antitumor activity of tazemetostat in population with tumors with aberrations in EZH2 or SWI/SNF complex pathways | Up to 2 years
  Molecular and clinical predictors of clinical outcomes will be investigated using logistic regression and Cox proportional hazards models. Potential predictors include clinical predictors and molecular correlates. Descriptive statistics and plotting of data will also be used to better understand potential relationships. All analyses will be considered exploratory and inference will be performed with appropriate caution.
Objective confirmed response | Up to 2 years
  Response will be assessed using the Response Evaluation Criteria in Solid Tumors (RECIST) criteria 1.1
Duration of response | Up to 2 years
  Response will be assessed using the RECIST criteria 1.1.
Best response | Up to 2 years
  Response will be assessed using the RECIST criteria 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Renouf, Principal Investigator — University Health Network Princess Margaret Cancer Center LAO
Locations (1):
- Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland, United States